CLINICAL TRIAL: NCT06733298
Title: Open-Label, Non-Randomized Study Investigating the Excretion Balance, Pharmacokinetics, and Metabolism of a Single Oral Dose of [14C]-Labeled RO7269162 in Healthy Male Participants
Brief Title: A Study Investigating [14C]-Labeled RO7269162 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP45325
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants will receive one oral dose of [14C]-labeled RO7269162 on Day 1.
  Interventions: Drug: [ 14C]-labeled RO7269162

INTERVENTIONS:
Drug: [ 14C]-labeled RO7269162 — Participants will receive one oral dose of [14C]-labeled RO7269162.

SUMMARY:
This study will investigate how RO7269162 labeled with a carbon tracer ([14C]) is absorbed, metabolized, and eliminated by the body after a single dose in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 35 to 64 years of age (inclusive), at screening
* Body weight ≥ 50 kg and body mass index within the range 18 to 30 kg/m2 (inclusive), at screening
* Male participants who, for 3 months after dosing of [14C]-RO7269162, agree to: remain abstinent (refrain from heterosexual intercourse) or use contraception as defined by the protocol with a partner that is a woman of childbearing potential; remain abstinent or use contraception with a pregnant female partner; refrain from donating sperm

Exclusion Criteria:

* History or evidence of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological, or allergic disease, metabolic disorder, cancer, or cirrhosis
* Any disease or condition that could interfere with the conduct of the study or pose an unacceptable risk to the participant
* History or evidence of any medical condition that could potentially alter the absorption, metabolism, or elimination of drugs
* Surgical history of the gastrointestinal (GI) tract affecting gastric motility or altering the GI tract (with the exception of uncomplicated appendectomy and hernia repair)
* History of malignancy
* Use of any prescription drugs, herbal supplements, and/or over-the-counter medication (OTC), dietary supplements (vitamins included) within 2 weeks before Day 1. Use of any prohibited food before study start and during the study as defined by the protocol
* Likely to need medication during the study period except for those defined by the protocol
* Are currently enrolled in, have participated in, or plan to participate in any other clinical study involving an investigational medicinal product or medical device study from within the 30 days directly preceding screening or within 5 times the elimination half-life, if known (whichever is longer), until completion of the follow-up visit
* Evidence of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Donation of blood or blood products for transfusion over 100 mL or significant blood loss within 2 months prior to screening through study completion, clinic discharge or early termination, inclusive. Donation of blood or plasma is not allowed throughout the entire study. Receipt of blood products within 2 months prior to Day -1 is not allowed
* Clinically significant history of hypersensitivity or allergic reactions
* Regular work with ionizing radiation or radioactive material, or exposure to ionizing radiation within 1 year prior to study drug administration

Ages: 35 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
[14C] recovery in urine | Up to Day 22 or Day 37
[14C] recovery in feces | Up to Day 22 or Day 37
Concentration of [14C] in whole blood | Up to Day 22 or Day 37
Plasma concentration of [14C] | Up to Day 22 or Day 37
Plasma concentration of RO7269162 | Up to Day 22 or Day 37
Amount of RO7269162 excreted in urine | Up to Day 22 or Day 37

SECONDARY OUTCOMES:
Amount of RO7269162 metabolites in plasma | Up to Day 22 or Day 37
Amount of RO7269162 metabolites in blood | Up to Day 22 or Day 37
Amount of RO7269162 metabolites excreted in urine | Up to Day 22 or Day 37
Amount of RO7269162 metabolites excreted in feces | Up to Day 22 or Day 37
Incidence and severity of adverse events | Up to Day 22 or Day 37

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- ICON Health sciences research center, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No